CLINICAL TRIAL: NCT00364741
Title: PeRioperative OXygen Fraction - Effect on Surgical Site Infection and Pulmonary Complications After Abdominal Surgery (The PROXI-trial)
Brief Title: Supplemental Oxygen and Complications After Abdominal Surgery (The PROXI-trial)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Danish Medical Research Council (Other)
Responsible Party: Lars S. Rasmussen, Department of Anaesthesia, HOC, Copenhagen University Hospital, Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2006-001710-32; GCP-2006-101; KF 02 306766
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Laparotomy
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Fraction of inspired oxygen (FiO2) = 0.30
  Interventions: Drug: Oxygen
- B (Active Comparator): FiO2 = 0.80
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — During and 2 hours after surgery

SUMMARY:
Aim: To investigate the effect of high intra- and postoperative oxygen concentration (80%, as opposed to normally 30%) on surgical wound infection and pulmonary complications after abdominal surgery.

Background: Surgical wound infection is a common and serious complication. Tissue oxygen tension is often low after surgery and the resistance against infection depends on this factor through bacterial killing by neutrophils. Oxygen is a substrate in this reaction, and it is hypothesized that by increasing the arterial oxygen tension, the risk of surgical wound infection is reduced. Previous studies to test this hypothesis have shown entirely different results. Hence, the clinical decision between high and normal oxygen concentration is still controversial.

Primary hypothesis of study: Use of 80% oxygen decreases the incidence of surgical wound infection after abdominal surgery.

Secondary objectives: To investigate the effect 80% oxygen on pulmonary complications (atelectasis, pneumonia, respiratory insufficiency), second operation, mortality and length of postoperative hospitalization and admission to intensive care unit after abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Laparotomy, acute or elective. In case of gynaecological surgery only if malignancy is suspected (defined as risk of ovarian malignancy index >200 or a specimen with atypical or neoplastic cells).

Exclusion Criteria:

* Other surgery within 30 days (except surgery in local anaesthesia).
* Chemotherapy within 3 months.
* Inability to give informed consent.
* Inability to keep oxygen saturation above 90% without supplemental oxygen (measured preoperatively by pulse oximetry).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Surgical wound infection | 14 days after surgery

SECONDARY OUTCOMES:
Atelectasis, pneumonia, respiratory insufficiency, second operation, mortality, length of postoperative hospitalization, admission to intensive care unit. | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lars S. Rasmussen, MD,DMSc,PHD, Study Chair — Dept. of Anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark; Jørn Wetterslev, MD, PHD, Study Director — Copenhagen Trial Unit, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark; Lars N. Jørgensen, MD, DMSc, Study Director — Dept. of Surgery, Copenhagen University Hospital, Bispebjerg, Copenhagen, Denmark; Christian S. Meyhoff, MD, PhD, Principal Investigator — Dept. of Anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark
Locations (14):
- Denmark (14):
  - Aarhus Sygehus, Aarhus
  - Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Copenhagen University Hospital, Amager, Copenhagen
  - Copenhagen University Hospital, Bispebjerg, Copenhagen
  - Copenhagen University Hospital, Gentofte, Hellerup
  - Copenhagen University Hospital, Herlev, Herlev
  - Holbaek Hospital, Holbæk
  - Kolding Hospital, Kolding
  - Nykoebing Falster Hospital, Nykoebing Falster
  - Naestved Hospital, Næstved
  - Slagelse Hospital, Slagelse
  - Funen County Hospital, Svendborg
  - Vejle Hospital, Vejle
  - Viborg Hospital, Viborg

REFERENCES:
- [Background] Meyhoff CS, Wetterslev J, Jorgensen LN, Henneberg SW, Simonsen I, Pulawska T, Walker LR, Skovgaard N, Helto K, Gocht-Jensen P, Carlsson PS, Rask H, Karim S, Carlsen CG, Jensen FS, Rasmussen LS; PROXI Trial Group. Perioperative oxygen fraction - effect on surgical site infection and pulmonary complications after abdominal surgery: a randomized clinical trial. Rationale and design of the PROXI-Trial. Trials. 2008 Oct 22;9:58. doi: 10.1186/1745-6215-9-58. PMID 18945347
- [Result] Meyhoff CS, Wetterslev J, Jorgensen LN, Henneberg SW, Hogdall C, Lundvall L, Svendsen PE, Mollerup H, Lunn TH, Simonsen I, Martinsen KR, Pulawska T, Bundgaard L, Bugge L, Hansen EG, Riber C, Gocht-Jensen P, Walker LR, Bendtsen A, Johansson G, Skovgaard N, Helto K, Poukinski A, Korshin A, Walli A, Bulut M, Carlsson PS, Rodt SA, Lundbech LB, Rask H, Buch N, Perdawid SK, Reza J, Jensen KV, Carlsen CG, Jensen FS, Rasmussen LS; PROXI Trial Group. Effect of high perioperative oxygen fraction on surgical site infection and pulmonary complications after abdominal surgery: the PROXI randomized clinical trial. JAMA. 2009 Oct 14;302(14):1543-50. doi: 10.1001/jama.2009.1452. PMID 19826023